CLINICAL TRIAL: NCT06963372
Title: Assessment of Health Effects of Air Purifier Interventions on Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Hwan-Cheol Kim, Professor, Inha University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-03-023
Record Dates: First submitted 2024-08-22; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases; Particulate Matter
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: A randomized, single-blind, crossover study was conducted at two university hospitals in Seoul and Incheon, involving 24 CKD patients and 24 healthy controls. Participants underwent two repeated measures with each receiving either a true filter or a sham filter in air purifiers for four weeks, separated by a two-week washout period. The sequence of filter application was counterbalanced between two groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A used an air purifier equipped with a true filter for four weeks, followed by a two-week washout period, and then used an air purifier with a sham filter.
  Interventions: Device: True filter (4w) → Washout (2w) → Sham filter (4w)
- Group B (Experimental): Group B used an air purifier equipped with a sham filter for four weeks, followed by a two-week washout period, and then used an air purifier with a true filter.
  Interventions: Device: Sham filter (4w) → Washout (2w) → True filter (4w)

INTERVENTIONS:
Device: True filter (4w) → Washout (2w) → Sham filter (4w) — Used a true filter for 4 weeks, followed by a 2-week washout, then used a sham filter for 4 weeks.
  Arms: Group A
Device: Sham filter (4w) → Washout (2w) → True filter (4w) — Used a sham filter for 4 weeks, followed by a 2-week washout, then used a true filter for 4 weeks.
  Arms: Group B

SUMMARY:
This exploratory study investigates the impact of indoor air quality improvement via air purifiers on the health of chronic kidney disease (CKD) patients.

A randomized, single-blind, crossover study with 24 CKD patients and 24 healthy controls was conducted at two hospitals. Participants used either a true filter or a sham filter in air purifiers for four weeks each, with a two-week washout period. True filters significantly reduced indoor PM2.5 levels compared to sham filters. Higher indoor PM2.5 levels were associated with increased cytokines (IL-1beta, IL-6, IL-8/CXCL8) and decreased hemoglobin, with ESR and PWV showing an increasing trend, particularly in CKD patients. True filters significantly reduced IL-1beta and IL-8/CXCL8 levels, with a borderline significant reduction in ABI. The study confirmed limited but notable effects of air purifiers on reducing PM2.5 and improving some health markers in CKD patients.

DETAILED DESCRIPTION:
Objectives:

Recent research has demonstrated that increasing levels of fine particulate matter (PM2.5) are associated with reduced glomerular filtration rates and elevated risks of chronic kidney disease (CKD) and end-stage renal disease (ESRD). To mitigate health impacts from PM2.5 exposure, recommendations include limiting outdoor activities, using air purifiers to improve indoor air quality, and wearing protective masks when outdoors. However, scientific evidence on the effectiveness of these interventions remains insufficient, particularly concerning how PM2.5 mitigation affects CKD progression. Therefore, this exploratory study aims to evaluate the impact of indoor air quality improvement via air purifiers on the health of CKD patients.

Methods:

A randomized, single-blind, crossover study was conducted at two university hospitals in Seoul and Incheon, involving 24 CKD patients and 24 healthy controls. Participants underwent two repeated measures with each receiving either a true filter or a sham filter in air purifiers for four weeks, separated by a two-week washout period. The sequence of filter application was counterbalanced between two groups. Data collection included surveys on lifestyle, medical history, and living environment, as well as blood, urine, and vascular endothelial function tests. The relationship between air purifier usage and health outcomes was analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient Group: Patients aged 20 years or older with stage 3 or higher chronic kidney disease (estimated glomerular filtration rate [eGFR] <60 mL/min/1.73 m²).
2. Control Group: Individuals aged 20 years or older who have not been told of any kidney function abnormalities based on blood tests within the past year and have never been diagnosed with chronic kidney disease. Baseline labs will be conducted, and only those with an eGFR ≥60 mL/min/1.73 m² will be enrolled. This group includes household members of the patient group or other healthy individuals.
3. Individuals who are not currently using a household air purifier.
4. Individuals who have consented to participate in the clinical study.

Exclusion Criteria:

1. Patients with stage 5 chronic kidney disease.
2. Individuals with a history of chronic obstructive pulmonary disease (COPD), asthma, allergy, cerebrovascular accident (CVA), malignancy (cancer), cardiovascular interventions, or those with an active infection.
3. Individuals taking immunosuppressive medications.
4. Patients with diabetes or hypertension whose blood sugar and blood pressure are uncontrolled (HbA1c > 8%, office SBP > 150 mmHg).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
IL-1beta in pg/mL | 0 weeks, 4 weeks, 6 weeks, 10 weeks
  Blood samples were collected to analyze cytokines.
IL-6 in pg/mL | 0 weeks, 4 weeks, 6 weeks, 10 weeks
  Blood samples were collected to analyze cytokines.
IL-8/CXCL8 in pg/mL | 0 weeks, 4 weeks, 6 weeks, 10 weeks
  Blood samples were collected to analyze cytokines.
IL-10 in pg/mL | 0 weeks, 4 weeks, 6 weeks, 10 weeks
  Blood samples were collected to analyze cytokines.
IFN-gamma in pg/mL | 0 weeks, 4 weeks, 6 weeks, 10 weeks
  Blood samples were collected to analyze cytokines.
TNF-alpha in pg/mL | 0 weeks, 4 weeks, 6 weeks, 10 weeks
  Blood samples were collected to analyze cytokines.

SECONDARY OUTCOMES:
Bood pressure (Systolic) in mmHg | 0 weeks, 4 weeks, 6 weeks, 10 weeks
Bood pressure (Diastolic) in mmHg | 0 weeks, 4 weeks, 6 weeks, 10 weeks
Pulse Wave Velocity in m/sec | 0 weeks, 4 weeks, 6 weeks, 10 weeks
  Pulse Wave Velocity in m/sec
Ankle-Brachial Pressure Index | 0 weeks, 4 weeks, 6 weeks, 10 weeks
  Ankle-Brachial Pressure Index (unitless)

CONTACTS AND LOCATIONS:
Overall Officials: Hwan-Cheol Kim, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No